CLINICAL TRIAL: NCT03681418
Title: Role of Ultrasound-Guided Lymph Node Biopsy in Axillary Staging of Breast Cancer.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mai El-Moataz Bellah Mohamed El-Sadek Khedrawy, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LNs Staging of Breast cancer
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
Keywords: Axillary Lymph Node Biopsy in Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with operable breast cancer (Other): Ultrasound-guided axillary lymph nodes FNAC and\or CNB.
  Interventions: Procedure: Ultrasound-guided axillary lymph nodes FNAC and\or CNB.

INTERVENTIONS:
Procedure: Ultrasound-guided axillary lymph nodes FNAC and\or CNB. — Ultrasound-guided axillary lymph node fine needle aspiration and\or core needle biopsy of the most suspicious lymph node. If all the lymph nodes appeared similar or normal, the lymph node that is lowest in the axilla will be selected because it is considered to most likely be the sentinel node.

SUMMARY:
The purpose of the study is to estimate the diagnostic accuracy of preoperative ultrasound-guided axillary lymph node biopsy for staging in patients with newly diagnosed breast cancer, and also to compare between ultrasound-guided fine needle aspiration cytology and core needle biopsy in their ability to detect metastatic disease in the axillary lymph nodes of patients with breast cancer.

DETAILED DESCRIPTION:
Axillary lymph node status is an extremely important prognostic factor in the assessment and treatment evaluation of patients with newly diagnosed breast cancer. Historically, axillary lymph node dissection (ALND) has been the reference standard for diagnosis and staging. However, this procedure can cause numerous postoperative problems, such as lymphedema , pain, impaired shoulder mobility and arm weakness. Furthermore, in this era of mammographic screening, axillary lymph node dissection yields negative results in 80%-85% of patients with T1 cancer.

Therefore, in recent years, sentinel lymph node biopsy (SNB) has replaced axillary dissection for lymph node staging at major medical centers. However, there are some practical issues to be resolved. For example, radiotracer distribution can be slow or faulty, valuable operating room time is expended, and pathologists must make quick decisions based on the analysis of frozen sections or there is the need to undergo two surgical interventions (i.e., removal of primary tumor and SNB, and in a next step completion ALND). If nodal positivity could be proven and documented preoperatively, sentinel lymph node biopsy could be bypassed and a decision will be made to perform axillary dissection, which is the standard of care in most node-positive patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with operable breast cancer regardless of whether lymph nodes are suspicious or not.

Exclusion Criteria:

* Patients who had previously undergone axillary surgery.
* Patients with metastatic disease and not planned for axillary surgery.
* Patients with a preoperative diagnosis of a benign lesion or ductal carcinoma in situ.
* Patients with severe uncorrectable bleeding diathesis.
* Patients refused to sign consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of preoperative ultrasound-guided axillary lymph node biopsy for staging in patients with newly diagnosed breast cancer. | Baseline.
  Accuracy will be determined by comparing the results of ultrasound-guided axillary lymph node biopsy to the gold standard which is the final pathological results from sentinel lymphadenectomy or axillary lymph node dissection.

SECONDARY OUTCOMES:
Accuracy of ultrasound-guided fine needle aspiration cytology and core needle biopsy in their ability to detect metastatic disease in the axillary lymph nodes of patients with a recent diagnosis of ipsilateral breast cancer. | Baseline.
  Ultrasound-guided fine needle aspiration and\or core needle biopsy of axillary lymph node of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Mai M. Khedrawy, M.B.B.CH, Principal Investigator — Assiut University; Hassan I. Metgally, professor, Study Director — Assiut University; Momtaz T. Allam, Lecturer, Study Director — Assiut University

REFERENCES:
- [Background] Swenson KK, Nissen MJ, Ceronsky C, Swenson L, Lee MW, Tuttle TM. Comparison of side effects between sentinel lymph node and axillary lymph node dissection for breast cancer. Ann Surg Oncol. 2002 Oct;9(8):745-53. doi: 10.1007/BF02574496. PMID 12374657
- [Background] Kumar R, Jana S, Heiba SI, Dakhel M, Axelrod D, Siegel B, Bernik S, Mills C, Wallack M, Abdel-Dayem HM. Retrospective analysis of sentinel node localization in multifocal, multicentric, palpable, or nonpalpable breast cancer. J Nucl Med. 2003 Jan;44(1):7-10. PMID 12515869
- [Background] Mainiero MB, Cinelli CM, Koelliker SL, Graves TA, Chung MA. Axillary ultrasound and fine-needle aspiration in the preoperative evaluation of the breast cancer patient: an algorithm based on tumor size and lymph node appearance. AJR Am J Roentgenol. 2010 Nov;195(5):1261-7. doi: 10.2214/AJR.10.4414. PMID 20966338